CLINICAL TRIAL: NCT01848561
Title: A Long-Term Non-Interventional Postmarketing Study to Assess Safety and Effectiveness of HUMIRA® (Adalimumab) in Patients With Moderately to Severely Active Ulcerative Colitis (UC)
Brief Title: A Long-Term Registry of Humira® (Adalimumab) in Patients With Moderately to Severely Active Ulcerative Colitis (UC)
Acronym: LEGACY
Status: Active, not recruiting | Type: Observational
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Other Study IDs: P11-282
Record Dates: First submitted 2013-05-03; First posted 2013-05-07 (Estimated); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Ulcerative Colitis (UC)
Keywords: Ulcerative Colitis; Registry; Adalimumab; Colitis; Gastroenteritis; Inflammatory Bowel Diseases; Gastrointestinal Diseases
MeSH Terms: conditions — Colitis, Ulcerative; Colitis; Gastroenteritis; Inflammatory Bowel Diseases; Gastrointestinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Immunomodulatory Therapy: Patients who are being prescribed and treated with Immunomodulatory Therapy
- Adalimumab (Humira) Treatment: Patients who are prescribed and treated with Adalimumab

SUMMARY:
This is a registry study to evaluate the long-term safety and effectiveness of adalimumab in patients with moderately to severely active UC who are treated as recommended in the product label.

ELIGIBILITY:
Inclusion Criteria:

* For enrollment into the HUMIRA treatment group; adult patients with moderately to severely active UC who has been prescribed HUMIRA therapy according to routine clinical practice and meets one of the following:

  1. Is currently taking HUMIRA therapy and has received at least 8 weeks of therapy; OR
  2. Is entering after participation in an Abbott or AbbVie sponsored UC study and; has received continuous HUMIRA therapy since initiation of therapy
* For enrollment into the IMM treatment group; adult patients with moderately to severely active UC who has been prescribed IMM therapy, is currently taking IMM therapy, and has received at least 12 consecutive weeks of IMM therapy
* Patients capable of and willing to grant authorization for use/disclosure of data being collected and provided to AbbVie prior to any registry-related data being collected, and to comply with the requirements of the Registry protocol

Exclusion Criteria:

* Patients on IMM therapy without a concurrent biologic if they cannot continue to be treated with IMM therapy or
* Patients who are being treated with any investigational agents and/or approved biologics other than Humira.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with moderately to severely active Ulcerative Colitis (UC) who have been prescribed HUMIRA according to the local label and adult patients being prescribed and treated with IMM (6-mercaptopurine or azathioprine) with no concurrent biologic use.
Sampling Method: Probability Sample
Enrollment: 8250 (Estimated)
Dates: Start 2013-04-29 (Actual); Primary Completion 2028-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of long term safety of Adalimumab in patients with moderately to severely active UC | 10 years observational period

SECONDARY OUTCOMES:
Evaluation of long term effectiveness of Adalimumab in patients with moderately to severely active UC who have had an inadequate response to conventional therapy | 10 years observational period

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (512):
- United States (169):
  - Birmingham Gastroenterology Associates P.C /ID# 102063, Birmingham, Alabama
  - University of Alabama at Birmingham - Main /ID# 131646, Birmingham, Alabama
  - Longwood Research /ID# 118662, Huntsville, Alabama
  - East View Medical Research, LLC /ID# 116259, Mobile, Alabama
  - Mobile Medical & Diagnostic Center, AL /ID# 102064, Mobile, Alabama
  - HOPE Research Institute /ID# 127947, Phoenix, Arizona
  - Duplicate_University of Arizona Cancer Center - North Campus /ID# 140387, Tucson, Arizona
  - University Of Arizona /ID# 117836, Tucson, Arizona
  - Arkansas Gastroenterology /ID# 113898, North Little Rock, Arkansas
  - Southern California Res. Ctr. /ID# 116898, Coronado, California
  - Moores Cancer Center at UC San Diego /ID# 133722, La Jolla, California
  - McGuire, Jr. La Mirada, CA /ID# 116257, La Mirada, California
  - Atay, Los Alamitos, CA /ID# 110175, Los Alamitos, California
  - Temecula Valley Endoscopy Ctr /ID# 118660, Murrieta, California
  - Community Clinical Trials, CA /ID# 117335, Orange, California
  - Digestive Care Medical Center /ID# 122075, San Carlos, California
  - Precision Research Institute - San Diego /ID# 103638, San Diego, California
  - Precision Research Institute - San Diego /ID# 113445, San Diego, California
  - Santa Monica Research Institut /ID# 118675, Santa Monica, California
  - Duplicate_St. Joseph Heritage Group - Yorba Linda /ID# 133721, Yorba Linda, California
  - Duplicate_Western States Clinical Research, Inc. /ID# 116237, Wheat Ridge, Colorado
  - Gastro Assoc of Fair County /ID# 113443, Bridgeport, Connecticut
  - Gastroenterology Center of Connecticut /ID# 102057, Hamden, Connecticut
  - Middlesex Hospital /ID# 122077, Middletown, Connecticut
  - Yale Univ Digestive Diseases /ID# 141987, New Haven, Connecticut
  - Georgetown University Hospital /ID# 113437, Washington D.C., District of Columbia
  - Brandon Premier Health Care, PA/Gulf Coast Research Group, LLC /ID# 148230, Brandon, Florida
  - Sarkis Clinical Trials /ID# 137948, Gainesville, Florida
  - Hollywood Research Center /Id# 214723, Hollywood, Florida
  - Ctr for Advanced Gastroenterol /ID# 116236, Maitland, Florida
  - Research Associates of South Florida,LLC /ID# 148212, Miami, Florida
  - Paradise Clnical Research, LLC /ID# 212027, Miami, Florida
  - Duplicate_Abel & Buchheim, P.R., Inc. /ID# 143863, Miami, Florida
  - Gastroenterology Group Naples /ID# 105837, Naples, Florida
  - Advanced Research Institute, Inc /ID# 211335, New Port Richey, Florida
  - Duplicate_North Florida Gastro Research /ID# 128538, Orange Park, Florida
  - Advent Health /ID# 145705, Orlando, Florida
  - Endoscopic Research, Inc. /ID# 136883, Orlando, Florida
  - Duplicate_Combined Research Orlando - Phase I-IV /ID# 141660, Orlando, Florida
  - Digestive Diseases Center /ID# 118116, Panama City, Florida
  - Palekar. Parkland, FL /ID# 108202, Parkland, Florida
  - BRCR Medical Center Inc /ID# 152015, Plantation, Florida
  - Advanced Medical Research Center /ID# 116235, Port Orange, Florida
  - Precision Clinical Research /ID# 127849, Sunrise, Florida
  - Digestive Disease Clinic /ID# 107162, Tallahassee, Florida
  - University of South Florida- Neuroscience Institute /ID# 213305, Tampa, Florida
  - Guardian Angels Health Center /ID# 209706, Tampa, Florida
  - South Florida Ctr Gastro, P.A. /ID# 166784, Wellington, Florida
  - Shafran Gastroenterology Ctr /ID# 117839, Winter Park, Florida
  - Winship Cancer Institute of Emory University /ID# 133724, Atlanta, Georgia
  - Atlanta Gastro Assoc /ID# 107164, Atlanta, Georgia
  - Gastroenterology Associates of Central Georgia, LLC /ID# 117838, Macon, Georgia
  - Atlanta Gastroenterology Spec /ID# 103619, Suwanee, Georgia
  - Grand Teton Research Group /ID# 108197, Idaho Falls, Idaho
  - Northwest Gastro, S.C. /ID# 103620, Arlington Heights, Illinois
  - Northwest Gastro, S.C. /ID# 145707, Arlington Heights, Illinois
  - Christie Clinic, LLC /ID# 116258, Champaign, Illinois
  - Northwestern University Feinberg School of Medicine /ID# 126760, Chicago, Illinois
  - Rush University Medical Center /ID# 132979, Chicago, Illinois
  - The University of Chicago Medical Center /ID# 114115, Chicago, Illinois
  - Duplicate_NorthShore University HealthSystem /ID# 107165, Evanston, Illinois
  - DM Clinical Research/Southwest /ID# 120635, Oak Lawn, Illinois
  - Duplicate_North Suburban Gastro Assoc /ID# 134437, Park Ridge, Illinois
  - Carle Foundation Hospital Digestive Health Research Center /ID# 117417, Urbana, Illinois
  - Iowa Digestive Disease Center - Clive /ID# 107159, Clive, Iowa
  - University of Iowa Hospitals and Clinics /ID# 134432, Iowa City, Iowa
  - University of Kansas Health Sy /ID# 134436, Kansas City, Kansas
  - Univ Kansas Med Ctr /ID# 120917, Kansas City, Kansas
  - Kansas Gasteroenterology /ID# 214827, Wichita, Kansas
  - Houma Digestive Health Special /ID# 125711, Houma, Louisiana
  - Gastro Clinic of Acadiana, LA /ID# 119155, Lafayette, Louisiana
  - Louisiana Research Center, LLC /ID# 102055, Shreveport, Louisiana
  - Investigative Clinical Research /ID# 102056, Annapolis, Maryland
  - University of Maryland, Baltimore /ID# 116897, Baltimore, Maryland
  - Duplicate_MGG Group Co, Inc.Chevy Chase Clinical Research /ID# 107157, Chevy Chase, Maryland
  - Gastro Center of Maryland /ID# 126969, Columbia, Maryland
  - Endoscopic Microsurgery Assoc /ID# 102065, Towson, Maryland
  - Attleboro Gastroenterology, PC /ID# 113899, Attleboro, Massachusetts
  - Commonwealth Clinical Studies /ID# 118597, Brockton, Massachusetts
  - University of Michigan Comprehensive Cancer Center Michigan Medicine /ID# 105836, Ann Arbor, Michigan
  - Huron Gastroenterology Assoc /ID# 132484, Ann Arbor, Michigan
  - Henry Ford Hospital /ID# 103617, Detroit, Michigan
  - Detroit Clinical Research Center /ID# 123235, Farmington Hills, Michigan
  - Mayo Clinic - Rochester /ID# 116899, Rochester, Minnesota
  - Univ of Mississippi Med Ctr,US /ID# 132981, Jackson, Mississippi
  - St. Louis University /ID# 163794, St Louis, Missouri
  - Washington University-School of Medicine /ID# 107156, St Louis, Missouri
  - CHI Health Research Center /ID# 116255, Omaha, Nebraska
  - Cooper Digestive Health Instit /ID# 103615, Mount Laurel, New Jersey
  - Duplicate_The Gastro Group of S. Jersey /ID# 129902, Vineland, New Jersey
  - Allied Gastrointestinal Associates /ID# 107158, Voorhees Township, New Jersey
  - NYU Langone Long Island Clinical Research Associates /ID# 107163, Lake Success, New York
  - Orlin & Cohen /ID# 117895, Lynbrook, New York
  - Progressive Gastroenterology Consultants /ID# 105835, Mineola, New York
  - Digestive Disease Care /ID# 133489, New Hyde Park, New York
  - North Shore University Hospital /ID# 127948, New Hyde Park, New York
  - Duplicate_Premier Medical Group /ID# 140388, New Windsor, New York
  - New York Gastroenterology Associates - Upper West Side /ID# 133689, New York, New York
  - The Mount Sinai Hospital /ID# 108201, New York, New York
  - Weill Cornell Medical College /ID# 135052, New York, New York
  - Manhattan Clinical Research, LLC /ID# 113442, New York, New York
  - Premier Medical Group - GI Division /ID# 140384, Poughkeepsie, New York
  - Gastoenterology Group of Rochester /ID# 113438, Rochester, New York
  - University of Rochester Medical Center /ID# 126152, Rochester, New York
  - Ctr Digest, Allergic & Imm Dis /ID# 125502, Williamsville, New York
  - Asheville Gastro Assoc /ID# 144367, Asheville, North Carolina
  - Cary Gastroenterology Assoc PA /ID# 108198, Cary, North Carolina
  - Univ NC Chapel Hill /ID# 102059, Chapel Hill, North Carolina
  - Atrium Health Carolinas Medical Center /ID# 126970, Charlotte, North Carolina
  - Charlotte Gastroenterology and Hepatology, PLLC /ID# 102058, Charlotte, North Carolina
  - Carolina Digestive Health Associates /ID# 108199, Charlotte, North Carolina
  - Carolinas Research center /ID# 211288, Charlotte, North Carolina
  - Atlantic Gastroenterology, PA /ID# 135536, Greenville, North Carolina
  - Carolina Research /ID# 134133, Greenville, North Carolina
  - Boice-Willis Clinic, P.A. /ID# 103618, Rocky Mount, North Carolina
  - Trial Management Associates /ID# 138459, Wilmington, North Carolina
  - Atrium Health Wake Forest Baptist Medical Center /ID# 113436, Winston-Salem, North Carolina
  - Cleveland Clinic Main Campus /ID# 108055, Cleveland, Ohio
  - Duplicate_Clinical Research Solutions /ID# 207698, Middleburg Heights, Ohio
  - ProMedica Physicians Digestive Healthcare /ID# 156529, Sylvania, Ohio
  - Avamar Center for Endoscopy /ID# 113440, Warren, Ohio
  - Southwoods Surgical Hospital /ID# 133038, Youngstown, Ohio
  - Northwest Gastroenterology Clinic /ID# 116896, Portland, Oregon
  - Penn State University and Milton S. Hershey Medical Center /ID# 133688, Hershey, Pennsylvania
  - Main Line Gastro Assoc /ID# 113446, Malvern, Pennsylvania
  - Drexel University /ID# 126968, Philadelphia, Pennsylvania
  - Duplicate_Temple University Hospital /ID# 108203, Philadelphia, Pennsylvania
  - Methodist Hospital /ID# 129461, Philadelphia, Pennsylvania
  - Guthrie Medical Group, PC /ID# 105838, Sayre, Pennsylvania
  - Duplicate_Bierwirth, Cranston, RI /ID# 113435, Cranston, Rhode Island
  - Medical University of South Carolina /ID# 113439, Charleston, South Carolina
  - Consultants in Gastroenterology - Columbia NE /ID# 126517, Columbia, South Carolina
  - Greenville Endoscopy Center /ID# 129900, Greenville, South Carolina
  - Biocentric Healthcare Research /ID# 213980, West Columbia, South Carolina
  - Rapid City Medical Center - GI Research /ID# 201191, Rapid City, South Dakota
  - Singaram Gastroenterology /ID# 113447, Sioux Falls, South Dakota
  - Erlanger Institute for Clinical Research /ID# 126151, Chattanooga, Tennessee
  - Duplicate_Franklin Endoscopy Center /ID# 113444, Franklin, Tennessee
  - Clinical Research Solutions /ID# 154153, Jackson, Tennessee
  - Mid-State Gastroenterology /ID# 125457, Murfreesboro, Tennessee
  - Baylor College of Medicine /ID# 103636, Houston, Texas
  - Duplicate_Kelsey-Seybold Clinic /ID# 125942, Houston, Texas
  - University of Texas MD Anderson Cancer Center /ID# 144198, Houston, Texas
  - Precision Research Institute, LLC /ID# 211340, Houston, Texas
  - Houston Digestive Dis Clinic /ID# 102076, Houston, Texas
  - Houston Endoscopy And Research Center - Katy Freeway /ID# 206978, Houston, Texas
  - Rio Grande Gastroenterology /ID# 210218, McAllen, Texas
  - Digestive Health Center /ID# 113897, Pasadena, Texas
  - Digestive Health Assoc of TX /ID# 116215, Plano, Texas
  - Gastroenterology Clinic of San /ID# 113441, San Antonio, Texas
  - San Antonio Gastro Assoc /ID# 143435, San Antonio, Texas
  - Baylor Scott & White Medical Center- Temple /ID# 103639, Temple, Texas
  - Digestive Health Spec of Tyler /ID# 138144, Tyler, Texas
  - Care Access - Ogden /ID# 213432, Ogden, Utah
  - Granger Medical Clinic /ID# 122896, West Valley City, Utah
  - University of Vermont Medical Center /ID# 102075, Burlington, Vermont
  - Gastro Assoc of Tidewater /ID# 102061, Chesapeake, Virginia
  - Gastro Assoc. of N. Va. /ID# 125495, Fairfax, Virginia
  - Emeritas Research Group, LLC /ID# 135537, Leesburg, Virginia
  - Digestive and Liver Disease Sp /ID# 125943, Norfolk, Virginia
  - Gastroenterology Ltd. /ID# 103640, Virginia Beach, Virginia
  - University of Washington /ID# 122076, Seattle, Washington
  - Confluence Health /ID# 118661, Wenatchee, Washington
  - Duplicate_Morgantown Surgical Associates /ID# 123082, Morgantown, West Virginia
  - St. Mary's Hospital /ID# 116915, Madison, Wisconsin
  - Univ of Wisconsin Hosp/Clinics /ID# 103637, Madison, Wisconsin
  - Wisconsin Center for Advanced Research /ID# 103616, Milwaukee, Wisconsin
  - Froedtert Memorial Lutheran Hospital /ID# 102066, Milwaukee, Wisconsin
  - Reach /Id# 116256, Monroe, Wisconsin
- Australia (14):
  - The Canberra Hospital /ID# 157980, Garran, Australian Capital Territory
  - Royal Prince Alfred Hospital /ID# 157986, Camperdown, New South Wales
  - Concord Repatriation General Hospital /ID# 157983, Concord, New South Wales
  - St Vincent's Hospital /ID# 157978, East Lismore, New South Wales
  - Hunter New England Local Health District /ID# 157999, New Lambton, New South Wales
  - Royal Brisbane and Women's Hospital /ID# 158086, Herston, Queensland
  - Mater Misericordiae Limited /ID# 164171, South Brisbane, Queensland
  - Royal Adelaide Hospital /ID# 158026, Adelaide, South Australia
  - Flinders Medical Centre /ID# 157979, Bedford Park, South Australia
  - Box Hill Hospital /ID# 157987, Box Hill, Victoria
  - Austin Health /ID# 157998, Heidelberg, Victoria
  - The Alfred Hospital /ID# 159261, Melbourne, Victoria
  - The Royal Melbourne Hospital /ID# 157993, Parkville, Victoria
  - Fiona Stanley Hospital /ID# 157992, Murdoch, Western Australia
- Austria (5):
  - Ordensklinikum Linz GmbH Elisabethinen /ID# 98555, Linz, Upper Austria
  - Klinik Landstrasse /ID# 121615, Vienna, Vienna
  - Duplicate_Medizinische Universitat Innsbruck,Universitatsklinik fur Innere Mediz /ID# 120775, Innsbruck
  - Krankenhaus der Barmherzigen Brueder Salzburg /ID# 120776, Salzburg
  - Landeskrankenhaus Salzburg-Universitaetsklinikum der PMU (LKH) /ID# 127897, Salzburg
- Belgium (15):
  - Duplicate_ZAS Vincentius /ID# 127398, Antwerp, Antwerpen
  - Duplicate_ZAS Middelheim /ID# 129116, Antwerp, Antwerpen
  - Imelda Ziekenhuis /ID# 127497, Bonheiden, Antwerpen
  - Universitair Ziekenhuis Antwerpen /ID# 142757, Edegem, Antwerpen
  - Sint-Trudo Ziekenhuis /ID# 127136, Sint-Truiden, Limburg
  - Onze Lieve Vrouw Hospital /ID# 127986, Aalst, Oost-Vlaanderen
  - AZ Sint-Lucas /ID# 127000, Ghent, Oost-Vlaanderen
  - UZ Gent /ID# 127985, Ghent, Oost-Vlaanderen
  - Vitaz /Id# 141601, Sint-Niklaas, Oost-Vlaanderen
  - Universitair Ziekenhuis Leuven /ID# 127984, Leuven, Vlaams-Brabant
  - AZ Maria Middelares /ID# 127489, Ghent
  - AZ Herentals /ID# 127135, Herentals
  - CHU de Liege /ID# 127983, Liège
  - Groupe Sante CHC - Clinique du MontLegia /ID# 127988, Liège
  - Duplicate_Clinical Saint-Luc Bouge /ID# 127987, Namur
- Canada (21):
  - GI Research & Associates /ID# 133723, Edmonton, Alberta
  - Duplicate_University of Alberta - Zeidler Ledcor Centre /ID# 144673, Edmonton, Alberta
  - Columbia Gastro Mgmnt Ltd /ID# 128719, New Westminster, British Columbia
  - Dr. M. Prest Inc. /ID# 134309, Surrey, British Columbia
  - Duplicate_University of British Columbia - Eye Care Centre, Vancouver General Ho /ID# 129995, Vancouver, British Columbia
  - Duplicate_(G.I.R.I.) GI Research Institute Foundation /ID# 129095, Vancouver, British Columbia
  - Percuro Clinical Research, Ltd /ID# 129996, Victoria, British Columbia
  - Dr. Everett Chalmers Reg Hosp. /ID# 135408, Fredericton, New Brunswick
  - Duplicate_QE II Health Sciences Centre /ID# 128916, Halifax, Nova Scotia
  - Bellini Medicine Professional /ID# 145706, Brampton, Ontario
  - Guelph GI and Surgery Clinic /ID# 128917, Guelph, Ontario
  - Charlton Medical Centre /ID# 135390, Hamilton, Ontario
  - Duplicate_University Hospital - London Health Sciences Centre /ID# 128915, London, Ontario
  - Lakeridge Health - Oshawa /ID# 128275, Oshawa, Ontario
  - Ottawa Hospital Research Institute /ID# 128918, Ottawa, Ontario
  - Hôpital Montfort /ID# 151588, Ottawa, Ontario
  - Kensington Screening Clinic /ID# 133720, Toronto, Ontario
  - CIUSSS de l'est de l'Ile-de-Montreal - Hopital Maisonneuve-Rosemont /ID# 130321, Montreal, Quebec
  - CHUM - Notre-Dame Hospital /ID# 151379, Montreal, Quebec
  - CIUSSS de l'Estrie - CHUS /ID# 133031, Sherbrooke, Quebec
  - Royal University Hospital /ID# 128720, Saskatoon, Saskatchewan
- Croatia (5):
  - Clinical Hospital Dubrava /ID# 127982, Zagreb, City of Zagreb
  - General Hospital Sveti Duh /ID# 127977, Zagreb, City of Zagreb
  - Duplicate_Klinicki bolnicki centar Osijek /ID# 127980, Osijek, County of Osijek-Baranja
  - Klinicki bolnicki centar Rijeka /ID# 127979, Rijeka, Primorje-Gorski Kotar County
  - Duplicate_Klinicki bolnicki centar Split /ID# 127978, Split, Split-Dalmatia County
- Denmark (4):
  - Rigshospitalet /ID# 98238, Copenhagen Ø, Capital Region
  - Herlev Hospital /ID# 98239, Herlev, Capital Region
  - Kobenhavns Universitet - Hvidovre Hospital (HH) /ID# 120557, Hvidovre, Capital Region
  - Aalborg University Hospital /ID# 119215, Aalborg, North Denmark
- France (27):
  - Chu de Nice-Hopital L'Archet Ii /Id# 98645, Nice, Alpes-Maritimes
  - CHU Clermont-Ferrand /ID# 98735, Clermont, Auvergne-Rhône-Alpes
  - Duplicate_CHU Hopital Nord /ID# 98639, Marseille, Bouches-du-Rhone
  - CHU Toulouse - Hopital Purpan /ID# 148183, Toulouse, Haute-Garonne
  - CHU Toulouse - Hopital Rangueil /ID# 147755, Toulouse, Haute-Garonne
  - CHU Montpellier - Hopital Saint Eloi /ID# 217142, Montpellier, Herault
  - CHU Grenoble - Hopital Michallon /ID# 98638, La Tronche, Isere
  - CHU Reims - Hôpital Robert Debre /ID# 98640, Reims, Marne
  - CHRU Nancy - Hopitaux de Brabois /ID# 127394, Vandœuvre-lès-Nancy, Meurthe-et-Moselle
  - Cabinet medical Dr ECUER /ID# 161671, Metz, Moselle
  - CHRU Lille - Hopital Claude Huriez /ID# 98737, Lille, Nord
  - Centre Hospitalier Universitaire de Saint Etienne - Hopital Nord /ID# 130978, St-Priest-en-Jarez, Pays de la Loire Region
  - HCL - Hopital Edouard Herriot /ID# 155711, Lyon, Rhone
  - HCL - Hopital Lyon Sud /ID# 98718, Pierre-Bénite, Rhone
  - GH Mutualiste Les Portes Du Sud /ID# 98722, Vénissieux, Rhone
  - CHU Amiens-Picardie Site Sud /ID# 98637, Amiens, Somme
  - Hospitalier Germon et Gauthier /ID# 137874, Béthune
  - Centre des consultations spécialisées de la sauvegarde /ID# 98719, Lyon
  - GHI Le Raincy - Montfermeil /ID# 98642, Montfermeil
  - Duplicate_APHP - Groupe Hospitalier 1 /ID# 98736, Paris
  - AP-HP - Hopital Saint-Antoine /ID# 141611, Paris
  - Duplicate_AP-HP - Hopital Cochin /ID# 98717, Paris
  - AP-HP - Hopital Bichat - Claude-Bernard /ID# 98641, Paris
  - Hôpital Charles-Nicolle /ID# 98721, Rouen
  - Cabinet Médical - Dr THEVENIN /ID# 98720, Saint-Quentin
  - Duplicate_Hopital Trousseau /ID# 98716, Tours
  - Hopital Beaujon /ID# 127395, Clichy, Île-de-France Region
- Germany (63):
  - Universitaetsklinikum Freiburg /ID# 98176, Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinik Heidelberg /ID# 98120, Heidelberg, Baden-Wurttemberg
  - Praxis Für Gastroent. Dr. Med. Lars Helmstädter, Prof. Dr. Med. Robert Ehehalt /ID# 125211, Heidelberg, Baden-Wurttemberg
  - Universitatsklinikum Mannheim /ID# 129279, Mannheim, Baden-Wurttemberg
  - Duplicate_Clinics of Sigmaringen /ID# 98216, Sigmaringen, Baden-Wurttemberg
  - Universitaetsklinikum Ulm /ID# 98202, Ulm, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen /ID# 128179, Erlangen, Bavaria
  - Internistisches Fachzentrum /ID# 123255, Memmingen, Bavaria
  - Duplicate_Isar Medizin Zentrum /ID# 125213, Munich, Bavaria
  - Duplicate_Gastroenterologie Im Josephinu /ID# 123496, Munich, Bavaria
  - Duplicate_LMU Klinikum Campus Grosshadern /ID# 98198, Munich, Bavaria
  - Innere Am Stadtpark /ID# 123015, Nuremberg, Bavaria
  - Mueller/Mueller-Ziehm, Hanover /ID# 130490, Hanover, Lower Saxony
  - Internistische Praxengemeinschaft Oldenburg /ID# 129120, Oldenburg, Lower Saxony
  - Gastroenterologische Gemeinschaftspraxis Stade /ID# 98206, Stade, Lower Saxony
  - Universitaetsmedizin Rostock /ID# 128396, Rostock, Mecklenburg-Vorpommern
  - Bank, Schwerin, DE /ID# 125215, Schwerin, Mecklenburg-Vorpommern
  - Klinikum Dortmund gGmbH /ID# 127061, Dortmund, North Rhine-Westphalia
  - Gastroenterologische Gemeinschaftspraxis Herne /ID# 98121, Herne, North Rhine-Westphalia
  - Gastroenterologische Gemeinschaftspraxis Minden /ID# 98115, Minden, North Rhine-Westphalia
  - Benner & Dommermuth /ID# 129119, Koblenz, Rhineland-Palatinate
  - Duplicate_St. Marien- und Annastiftskrankenhaus /ID# 98235, Ludwigshafen am Rhein, Rhineland-Palatinate
  - Eugastro /ID# 98178, Leipzig, Saxony
  - Universitaetsklinikum Leipzig /ID# 98116, Leipzig, Saxony
  - Internistische Gemienschaftspraxis fuer Verdauungs- und Stoffwechselerkrankungen /ID# 98119, Leipzig, Saxony
  - Private Practice - Dr. Thomas Zeisler /ID# 98218, Halle, Saxony-Anhalt
  - Krankenhaus Martha-Maria Halle-Doelau /ID# 122935, Halle, Saxony-Anhalt
  - Gastroenterologisch - Hepatologisches MVZ Kiel GmbH /ID# 127798, Kiel, Schleswig-Holstein
  - Universitaetsklinikum Jena /ID# 127496, Jena, Thuringia
  - Klinikum Altenburger Land /ID# 131748, Altenburg
  - Praxis Dres. Roesler und Lachma /ID# 128466, Bayreuth
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 129115, Berlin
  - Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 129117, Berlin
  - Duplicate_Charite Universitaetsmedizin Berlin - Campus Mitte /ID# 98124, Berlin
  - Gastroenterologische Spezialpraxis am Wittenbergplatz /ID# 98117, Berlin
  - Charite Universitaetsklinikum Berlin - Campus Benjamin Franklin /ID# 130318, Berlin
  - DRK Kliniken Berlin Westend /ID# 98179, Berlin
  - Krankenhaus Waldfriede /ID# 98200, Berlin-Zehlendorf
  - Klinikum Ruhr Univ Bochum /ID# 148107, Bochum
  - Stadtisches Klinikum Braunschweig /ID# 98123, Braunschweig
  - Universitaetsmedizin Essen St. Josef Krankenhaus Werden /ID# 98196, Essen
  - Klinikum Garmisch-Partenkirchen /ID# 127915, Garmisch-Partenkirchen
  - Asklepios Klinik St. Georg /ID# 125216, Hamburg
  - Forstep /ID# 125206, Hamburg
  - Magen-Darm-Zentrum /ID# 141610, Hamburg
  - Gastroenterologie Fontenay /ID# 98195, Hamburg
  - Israelitisches Krankenhaus Hamburg /ID# 98197, Hamburg
  - Asklepios Westklinikum Hamburg /ID# 127492, Hamburg
  - Duplicate_Gastroenterologie Studien -CED /ID# 98205, Hamburg
  - Graefin v.Waldersee&Partner, H /ID# 141607, Hamburg
  - Hoffstadt, Iserlohn, DE /ID# 98208, Iserlohn
  - Otto-von-Guericke-Universitaet /ID# 129227, Magdeburg
  - Medizinisches Versorgungszentrum Portal 10 /ID# 98122, Münster
  - Gastro Campus Research GbR /ID# 125558, Münster
  - Klinikum Neumarkt /ID# 123016, Neumarkt
  - Klinikum Nuernberg Nord /ID# 134976, Nuremberg
  - Universitaetsklinikum Regensburg /ID# 141606, Regensburg
  - Praxiszentrum Altemalzerei /ID# 129001, Regensburg
  - Biewer/Mohl, Saarbruecken, DE /ID# 98204, Saarbrücken
  - Ambulanzzentrum Schweinfurt /ID# 123238, Schweinfurt
  - Kardalinos, Stuhr, DE /ID# 98201, Stuhr
  - Internistische Praxisgemeinschaft /ID# 129000, Weyhe
  - Loehr, Wiesbaden, DE /ID# 98217, Wiesbaden
- Greece (11):
  - Hygeia Hospital /ID# 128637, Amaroussio, Attica
  - General Hospital of Athens Ippokratio /ID# 128638, Athens, Attica
  - General Hospital of Athens Laiko /ID# 129280, Athens, Attica
  - Iatriko Kentro Athinon /ID# 98762, Marousi, Attica
  - General University Hospital of Alexandroupolis /ID# 128636, Alexandroupoli
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 98756, Athens
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 98761, Athens
  - Venizeleio General Hospital /ID# 98757, Heraklion
  - University General Hospital of Ioannina /ID# 127390, Ioannina
  - Theageneio Anticancer Hospital /ID# 141670, Thessaloniki
  - General Hospital of Thessaloniki Hippokrateio /ID# 127400, Thessaloniki
- Ireland (7):
  - Connolly Hospital Blanchardstown /ID# 98895, Abbotstown, Dublin
  - Mater Misericordiae Univ Hospital /ID# 119054, Dublin, Dublin
  - St James Hospital /ID# 149406, Dublin, Dublin
  - St Vincent's University Hospital /ID# 116835, Elm Park, Dublin
  - Beaumont Hospital /ID# 98775, Dublin
  - Duplicate_Adelaide and Meath Hosp,IE /ID# 117947, Dublin
  - Duplicate_Galway University Hospital /ID# 98763, Galway
- Israel (10):
  - Meir Medical Center /ID# 129238, Kfar Saba, Central District
  - Yitzhak Shamir Medical Center /ID# 128996, Ẕerifin, Central District
  - Hillel Yaffe Medical Center /ID# 129047, Hadera, Haifa District
  - Shaare Zedek Medical Center /ID# 126638, Jerusalem, Jerusalem
  - Gastroenterology Institute, Division of Medicine /ID# 132530, Jerusalem, Jerusalem
  - Clalit Health Services /ID# 129237, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 129281, Ramat Gan, Tel Aviv
  - Rambam Health Care Campus /ID# 129282, Haifa
  - Zavulun Medical Centre /ID# 129048, Kiriat Bialik
  - Duplicate_Baruch-Padeh Poriya Medical /ID# 141671, Lower Galilee
- Italy (29):
  - Duplicate_IRCCS AOU di Bologna - Policlinico Sant'Orsola-Malpighi /ID# 137945, Bologna, Emilia-Romagna
  - Duplicate_Azienda Ospedaliero Universitaria Careggi /ID# 137946, Florence, Firenze
  - Fondazione di Religione e di Culto Casa Sollievo della Sofferenza /ID# 137939, San Giovanni Rotondo, Foggia
  - Ospedale San Martino /ID# 137947, Genoa, Genova
  - IRCCS Istituto Clinico Humanitas /ID# 141382, Rozzano, Lombardy
  - ASST Fatebenefratelli Sacco /ID# 137944, Milan, Milano
  - ASST Fatebenefratelli Sacco /ID# 141716, Milan, Milano
  - Azienda Ospedaliera Universitaria Federico II /ID# 141381, Naples, Napoli
  - Duplicate_Policlinico Universitario Campus Bio-Medico /ID# 141393, Rome, Roma
  - Azienda Ospedaliera Universitaria Policlinico Tor Vergata /ID# 145912, Rome, Roma
  - Azienda Ospedaliera San Camillo Forlanini /ID# 144211, Rome, Roma
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I /ID# 144080, Rome, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS-Università Cattolica /ID# 141396, Rome, Roma
  - A.O. Ordine Mauriziano di Torino /ID# 137942, Turin, Torino
  - IRCCS Ospedale Sacro Cuore Don Calabria /ID# 137940, Negrar, Verona
  - A.O.U. Consorziale Policlinico di Bari /ID# 144213, Bari
  - ASST degli Spedali Civili di Brescia /ID# 137943, Brescia
  - Duplicate_Fondazione Poliambulanza Istituto Ospedaliero /ID# 141593, Brescia
  - Ospedale Cannizzaro /ID# 138142, Catania
  - Congregazione delle Suore Infermiere dell'Addolorata - Ospedale Valduce /ID# 155712, Como
  - Azienda Ospedaliera Universitaria Gaetano Martino /ID# 144212, Messina
  - Policlinico San Donato /ID# 141383, Milan
  - Ospedale S Giuseppe /ID# 141395, Milan
  - Duplicate_Seconda Universita' di Napoli /ID# 141717, Naples
  - Azienda Ospedaliero Universitaria Maggiore della Carita di Novara /ID# 144084, Novara
  - Azienda Ospedale-Universita Padova /ID# 137941, Padua
  - Duplicate_Azienda Ospedaliera Universitaria Paolo Giaccone /ID# 141397, Palermo
  - Azienda Ospedaliera Ospedali Riuniti Villa Sofia Cervello /ID# 141392, Palermo
  - Duplicate_A.O. Circolo e Fondazione Macc /ID# 141394, Varese
- Mexico (13):
  - Morales Vargas Centro de Investigacion S.C. /ID# 131390, León, Guanajuato
  - Asociacion Mexicana para la Investigacion Clinica /ID# 128387, Pachuca, Hidalgo
  - Instituto de Salud Digestiva /ID# 157435, Guadalajara, Jalisco
  - Issste /Id# 128386, Guadalajara, Jalisco
  - Clinica de Investigacion en Reumatologia y Obesidad S.C. /ID# 129318, Guadalajara, Jalisco
  - Clinica de Higado & Gastroenterologia Integral SC /ID# 128376, Cuernavaca, Morelos
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez /ID# 128375, Monterrey, Nuevo León
  - Investigacion y Biomedicina de Chihuahua /ID# 150115, Chihuahua City
  - Torre de Especialidades Medica /ID# 154276, Metepec
  - Centro Especializado en Diabetes, Obesidad y Prevencion de Enfermedades Cardiova /ID# 138113, Mexico City
  - Umsi /Id# 149283, Mexico City
  - Ruiz Flores, Monterrey, MX /ID# 128379, Monterrey NL
  - Vega Fonseca, San Luis Potosi /ID# 128380, San Luis Potosí City
- Netherlands (8):
  - Zuyderland Medisch Centrum /ID# 98241, Heerlen, Limburg
  - Olvg /Id# 98336, Amsterdam, North Holland
  - Isala /ID# 98317, Zwolle, Overijssel
  - Leids Universitair Medisch Centrum /ID# 127402, Leiden, South Holland
  - Erasmus Medisch Centrum /ID# 98337, Rotterdam, South Holland
  - Franciscus Gasthuis & Vlietland, Locatie Gasthuis /ID# 127904, Rotterdam, South Holland
  - Meander Medisch Centrum /ID# 98338, Amersfoort, Utrecht
  - Rijnstate /ID# 127397, Arnhem
- Christchurch Hospital /ID# 164265, Christchurch, Canterbury, New Zealand
- Akershus Universitetssykehus_MAIN /ID# 127159, Lorenskog, Akershus, Norway
- Puerto Rico (4):
  - Perez Jimenz Gastroenterologo /ID# 110135, Mayagüez
  - Gastro-Hepato & Geriatric Ctr /ID# 113135, Ponce
  - Henry A. Rodriguez Ginorio, MD /ID# 113448, San Juan
  - School of Medicine University of Puerto Rico-Medical Science Campus /ID# 102067, San Juan
- Spain (69):
  - Complejo Hospitalario Universitario A Coruña /ID# 129002, A Coruña, A Coruna
  - Hospital Arquitecto Marcide - Complejo Hospitalario Universitario de Ferrol /ID# 129124, Ferrol, A Coruna
  - Complejo Hospitalario Universitario de Santiago (CHUS) /ID# 98619, Santiago de Compostela, A Coruna
  - Hospital General Universitario de Elche /ID# 129121, Elche, Alicante
  - Hospital Universitario San Juan de Alicante /ID# 130167, Sant Joan d'Alacant, Alicante
  - Hospital de Manacor /ID# 128348, Manacor, Balearic Islands
  - Hospital Universitari Son Espases /ID# 148214, Palma de Mallorca, Balearic Islands
  - Hospital Universitario Germans Trias i Pujol /ID# 98592, Badalona, Barcelona
  - Hospital Sant Joan de Deu /ID# 151342, Esplugues de Llobregat, Barcelona
  - Hospital Sant Joan de Deu /ID# 155774, Esplugues de Llobregat, Barcelona
  - Hospital Universitari de Bellvitge /ID# 98584, L'Hospitalet de Llobregat, Barcelona
  - Consorci Corporacio Sanitaria Parc Tauli Sabadell /ID# 98585, Sabadell, Barcelona
  - Hospital de Viladecans /ID# 155500, Viladecans, Barcelona
  - Duplicate_Hospital Universitario de Jerez de la Frontera /ID# 128345, Jerez de la Frontera, Cadiz
  - Hospital Universitario Marques de Valdecilla /ID# 98581, Santander, Cantabria
  - Hospital General de Castellon /ID# 128351, Castellon, Castellon
  - Hospital General La Mancha Centro /ID# 98588, Alcázar de San Juan, Ciudad Real
  - Hospital Universitario Reina Sofia /ID# 98586, Córdoba, Cordoba
  - Hospital Comarcal Santa Ana de Motril /ID# 129040, Motril, Granada
  - Hospital Alto Guadalquivir /ID# 129006, Andújar, Jaen
  - Hospital Universitario Dr. Negrin /ID# 98578, Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Principe de Asturias /ID# 131751, Alcalá de Henares, Madrid
  - Hospital Universitario Fundacion Alcorcon /ID# 98576, Alcorcón, Madrid
  - Hospital Universitario de Fuenlabrada /ID# 98591, Fuenlabrada, Madrid
  - Hospital General de Mostoles /ID# 130319, Móstoles, Madrid
  - Hospital Universitario Infanta Cristina /ID# 98635, Parla, Madrid
  - Hospital Infanta Sofia /ID# 98615, San Sebastián de los Reyes, Madrid
  - Hospital de Antequera /ID# 129041, Antequera, Malaga
  - Hospital General Universitario Santa Lucia /ID# 129125, Cartagena, Murcia
  - Complejo Hospitalario Universitario Ourense /ID# 128349, Ourense, Ourense
  - Hospital Xeral Cies (CHUVI) /ID# 129515, Vigo, Pontevedra
  - Hospital Meixoeiro (CHUVI) /ID# 128355, Vigo, Pontevedra
  - Hospital Universitario de Cabuenes /ID# 141998, Gijón, Principality of Asturias
  - Hospital Universitario Central de Asturias /ID# 98617, Oviedo, Principality of Asturias
  - Hospital Universitario Canarias /ID# 129037, San Cristóbal de La Laguna, Santa Cruz De Tenerife
  - Hospital de Sagunto /ID# 98587, Sagunto, Valencia
  - Hospital San Eloy /ID# 147830, Barakaldo, Vizcaya
  - Hospital Universitario Basurto /ID# 129123, Bilbao, Vizcaya
  - Hospital Universitario de Galdakao /ID# 98618, Galdakao, Vizcaya
  - Hospital General Universitario de Alicante Doctor Balmis /ID# 128467, Alicante
  - Hospital Parc de Salut del Mar /ID# 126637, Barcelona
  - Hospital de Sant Joan Despi Moises Broggi /ID# 128347, Barcelona
  - Hospital San Pedro de Alcantara /ID# 98579, Cáceres
  - Hospital Universitario de Girona Doctor Josep Trueta /ID# 130049, Girona
  - Duplicate_Hospital San Jorge Huesca /ID# 149628, Huesca
  - Hospital Universitario de Jaen /ID# 129035, Jaén
  - Hospital de Leon /ID# 131750, León
  - Hospital Universitario de la Princesa /ID# 98580, Madrid
  - Hospital General Universitario Gregorio Maranon /ID# 98558, Madrid
  - Hospital Universitario Ramon y Cajal /ID# 98596, Madrid
  - Hospital Clinico San Carlos /ID# 98577, Madrid
  - Hospital Universitario 12 de Octubre /ID# 98575, Madrid
  - Hospital Universitario La Paz /ID# 98582, Madrid
  - Hospital Universitario Virgen de la Victoria /ID# 129038, Málaga
  - Complejo Hospitalario Universitario de Pontevedra /ID# 128354, Pontevedra
  - Hospital Universitario de Salamanca /ID# 98589, Salamanca
  - Hospital General de Segovia /ID# 148926, Segovia
  - Hospital Universitario Virgen Macarena /ID# 128346, Seville
  - Hospital Universitario Virgen del Rocio /ID# 98557, Seville
  - Hospital Universitario Virgen de Valme /ID# 129036, Seville
  - Hospital Universitari Joan Xxiii De Tarragona /ID# 129122, Tarragona
  - Hospital Virgen de la Salud /ID# 98595, Toledo
  - Hospital Clinico Universitario de Valencia /ID# 131749, Valencia
  - Consorci Hospital General Universitario de Valencia /ID# 98616, Valencia
  - Hospital Universitario y Politecnico La Fe /ID# 98597, Valencia
  - Hospital Rio Hortega /ID# 98590, Valladolid
  - Hospital Clinico Universitario Lozano Blesa /ID# 98556, Zaragoza
  - Hospital Universitario Miguel Servet /ID# 131188, Zaragoza
  - Hospital Royo Villanova /ID# 149850, Zaragoza
- Sweden (7):
  - Karolinska University Hospital Solna /ID# 171247, Solna, Stockholm County
  - Capio St Gorans Sjukhus /ID# 126123, Stockholm, Stockholm County
  - Sodersjukhuset /ID# 124158, Stockholm, Stockholm County
  - Danderyd Hospital /ID# 98897, Stockholm, Stockholm County
  - Uppsala University Hospital /ID# 120558, Uppsala, Uppsala County
  - Duplicate_Sahlgrenska University Hospital /ID# 141672, Gothenburg, Västra Götaland County
  - Skaraborgs Sjukhus Skovde /ID# 98898, Skövde, Västra Götaland County
- United Kingdom (29):
  - Warrington and Halton Hospitals NHS Foundation Trust /ID# 144089, Warrington, Cheshire West And Chester
  - County Durham and Darlington NHS Foundation Trust /ID# 145914, Darlington, County Durham
  - Derriford Hospital and the Royal Eye Infirmary /ID# 157432, Plymouth, Devon
  - University Hospitals Dorset NHS Foundation Trust /ID# 164108, Poole, Dorset
  - Hull University Teaching Hospitals NHS Trust /ID# 98899, Hull, East Riding Of Yorkshire
  - Hammersmith Hospital /ID# 145916, London, England
  - Hampshire Hospitals NHS Foundation Trust /ID# 98900, Basingstoke, Essex
  - Gartnavel General Hospital /ID# 153818, Glasgow, Glasgow City
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 145703, London, Greater London
  - University Hospital Southampton NHS Foundation Trust /ID# 145676, Southampton, Hampshire
  - James Paget University Hospitals NHS Foundation Trust /ID# 164106, Great Yarmouth, Norfolk
  - The Queen Elizabeth Hospital, Kings Lynn NHS Foundation Trust /ID# 145937, Kings Lynn, Norfolk
  - Nottingham City Hospital /ID# 145678, Nottingham, Nottinghamshire
  - West Suffolk Hospital /ID# 164105, Bury St Edmunds, Suffolk
  - Kingston Hospital NHS Foundation Trust /ID# 164109, Kingston upon Thames, Surrey
  - UH Coventry & Warwickshire /ID# 145680, Coventry, Warwickshire
  - Leeds Teaching Hospitals NHS Trust /ID# 157949, Leeds, West Yorkshire
  - Blackpool Teaching Hospitals NHS Foundation Trust /ID# 164213, Blackpool
  - Duplicate_Cambridge University Hospitals NHS Foundation Trust /ID# 145704, Cambridge
  - The Dudley Group NHS Foundation Trust /ID# 164119, Dudley
  - Kaiser Perm Riverside Med Ctr /ID# 146043, Fontana
  - London North West University Healthcare NHS Trust /ID# 145953, Harrow
  - Isle of Wight NHS Trust /ID# 168166, Isle of Wight
  - King's College Hospital NHS Foundation Trust /ID# 145698, London
  - Manchester University NHS Foundation Trust /ID# 145702, Manchester
  - Stockport NHS foundation trust /ID# 144090, Stockport
  - The Royal Wolverhampton NHS Trust /ID# 164209, Wolverhampton
  - The Royal Wolverhampton NHS Trust /ID# 98901, Wolverhampton
  - Yeovil Hospital - Somerset NHS Foundation Trust) /ID# 146042, Yeovil

REFERENCES:
- See also: Related Info — http://www.rxabbvie.com